CLINICAL TRIAL: NCT00541411
Title: Phase II Pilot Study of Vincristine, Adriamycin, Actinomycin D, Ifosfamide Combination Chemotherapy in Ewing's Sarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2031-065
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Ewing's Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — IVA protocol

INTERVENTIONS:
Drug: Vincristine, Actinomycin-D, Ifosfamide — Chemotherapy

SUMMARY:
Phase II Pilot Study of Vincristine, Adriamycin, Actinomycin D, Ifosfamide combination chemotherapy in Ewing's Sarcoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ewing's Sarcoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2003-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | overall

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Memon, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia